CLINICAL TRIAL: NCT03796884
Title: Phase II Randomized, Placebo-Controlled Trial of Linaclotide to Demonstrate Bioactivity in Patients With Sporadic Colorectal Adenomas and With Colorectal Cancer
Brief Title: Linaclotide in Treating Patients With Stages 0-3 Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, scott waldman, Associate Professor, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18F.524; CDMRP-CA170223 (Other Grant/Funding Number: DOD); JT 13271 (Other: JeffTrial Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Adenoma; Stage 0 Colorectal Cancer AJCC v8; Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — linaclotide; Tyrosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (linaclotide) (Experimental): Patients receive linaclotide PO daily on days 1-7 and undergo standard of care colonoscopy or surgery on day 7.
  Interventions: Drug: Linaclotide
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-7 and undergo standard of care colonoscopy or surgery on day 7.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Linaclotide — Given PO
  Other Names: 851199-59-2; Linzess; [9-L-tyrosine]heat-stable enterotoxin (Escherichia coli)-(6-19)-peptide; L-Tyrosine; L-cysteinyl-L-cysteinyl-L-alpha-glutamyl-L-tyrosyl-L-cysteinyl-L-cysteinyl-L- asparaginyl-L-prolyl-L-alanyl-L-cysteinyl-L-threonylglycyl-L-cysteiny; cyclic (1->6), (2->10), (5->13)-tris(disulfide); MD-1100
  Arms: Arm I (linaclotide)
Other: Placebo — Given PO
  Arms: Arm II (placebo)

SUMMARY:
This phase II trial studies the how well linaclotide works in treating patients with stages 0-3 colorectal cancer. Linaclotide is a very small protein that binds to receptors on intestinal cells and makes them secrete water and salt.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether, compared to placebo, linaclotide administered as a single oral daily dose x 7 days, induces a pharmacodynamics (PD) effect on cGMP levels, based on biopsy samples of adenomas or resected colorectal adenocarcinomas.

SECONDARY OBJECTIVES:

I. To compare Ki-67, guanylin levels and GUCY2C expression in adenomas and cancers versus normal tissue after exposure to linaclotide or placebo.

II. To confirm the safety and tolerability of linaclotide in sporadic adenoma and cancer patients.

TRANSLATIONAL OBJECTIVE:

I. To assess the pharmacodynamic effect of linaclotide on pathway-specific biomarkers relevant to GUCY2C signaling (i.e. VASP phosphorylation), markers of mutant APC-beta-catenin signaling (beta-catenin levels, beta-catenin nuclear localization, axin levels, c-Myc levels, guanylin levels, PCNA expression), based on adenoma/cancer and normal mucosa biopsy samples obtained by endoscopy following linaclotide or placebo exposure.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive linaclotide orally (PO) daily on days 1-7 and undergo standard of care colonoscopy or surgery on day 7.

ARM II. Patients receive placebo PO QD on days 1-7 and undergo standard of care colonoscopy or surgery on day 7.

After completion of study treatment, patients are followed up at day 14.

ELIGIBILITY:
Inclusion Criteria:

* History of 1 or more sporadic colorectal adenoma on previous endoscopy (adenoma cohort) or stage 0-3 biopsy proven colorectal cancer (CRC) (colorectal cancer cohort) who are scheduled for a surgical procedure
* Ability to understand and willingness to sign a written informed consent document and follow study procedures
* Ability to swallow capsules without difficulty
* Ability to maintain pill diaries
* Willingness to employ adequate contraception for men and women of childbearing potential for the duration of the study. Acceptable methods include double barrier methods, intrauterine device (IUD), postmenopausal status, and/or documentation of surgical sterilization
* Participants must have no chronic, clinically severe health issues which, in the opinion of their physician or the research team, could preclude trial activities including the one week drug exposure phase

Exclusion Criteria:

* History of gastroparesis
* History of celiac disease
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Microscopic colitis, including collagenous colitis
* Has taken linaclotide within 30 days prior to consent
* Any malignancy except colorectal cancer or any active radiotherapy or cytotoxic chemotherapy within the last 6 months of baseline. Participants with a history of basal cell or squamous cell skin cancer may be enrolled at the discretion of the investigator
* Participants may not be receiving any other investigational agents, or be active participants in any clinical trials. If participants previously participated in a clinical trial, a 30 day washout period for the investigational drug is needed before the participant can be considered for this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to linaclotide
* Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or lactating women
* History of bleeding/coagulation problems. Concurrent use of nonsteroidal anti-inflammatory drugs (NSAIDs) including aspirin is acceptable
* Any medical condition judged by the investigator to constitute a risk to safe participation
* At risk for obstructing or near-obstructing mechanical gastrointestinal obstruction
* Chronic use of anti-coagulants or non-NSAID anti-platelet agents will serve as an exclusion only when such medications cannot be safely discontinued before study related endoscopy or surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics effect on cGMP levels | Up to 2 years, plus an additional 12 months for primary analysis
  Will compare cGMP levels in adenomas between study arms using a two-sample t-test (alpha=.05; two-sided) or Wilcoxon rank sum test.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From the time of first dose of linaclotide or placebo until resolution, if related to linaclotide, or through 30 days after occurrence
  All participants will be evaluated for toxicity. Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be used to summarize adverse events associated with linaclotide.
Ki-67 expression | Up to 2 years
  Wilcoxon rank sum test will be used to compare Ki-67 expression in adenomas across arms.
GUCY2C expression | Up to 2 years
  Wilcoxon rank sum and Fisher's exact tests will be used to compare GUCY2C expression between study arms.
Guanylin levels | Up to 2 years
  Wilcoxon rank sum and Fisher's exact tests will be used to compare guanylin levels between study arms.

OTHER OUTCOMES:
VASP serine 239 phosphorylation | Up to 2 years
  Assessed by immunoblot analysis. Wilcoxon rank sum and Fisher's exact tests will be used to compare VASP phosphorylation between study arms.
Beta-catenin levels | Up to 2 years
  Assessed by immunoblot analysis. Wilcoxon rank sum and Fisher's exact tests will be used to compare beta-catenin accumulation and downstream signaling between study arms.
Beta-catenin nuclear localization | Up to 2 years
  Assessed by immunofluorescence. Wilcoxon rank sum and Fisher's exact tests will be used to compare beta-catenin accumulation and downstream signaling between study arms
Axin and c-Myc messenger ribonucleic acid (mRNA) levels | Up to 2 years
  Assessed by quantitative reverse transcriptase-polymerase chain reaction. Wilcoxon rank sum and Fisher's exact tests will be used to compare axin and c-Myc mRNA levels between study arms.
PCNA expression | Up to 2 years
  Assessed by immunofluorescence.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Waldman, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (3):
- United States (3):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - VA Puget Sound Health Care Sysem, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Thomas Jefferson University Hospital — https://www.jeffersonhealth.org/locations/thomas-jefferson-university-hospital